CLINICAL TRIAL: NCT02125162
Title: A Single-dose, Randomized, 3-period, Crossover Study to Evaluate the Relative Bioavailability of BCX4161 Formulated as a Soft Gelatin Capsule to BCX4161 Formulated as a Hard Gelatin Capsule and the Effect of Food on BCX4161 Pharmacokinetics
Brief Title: A Study of the Relative Bioavailability of a New Formulation of BCX4161 and the Effect of Food on BCX4161
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BCX4161-104
Record Dates: First submitted 2014-04-24; First posted 2014-04-29 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Hereditary Angioedema
Keywords: BCX4161; BioCryst; hereditary angioedema; relative bioavailability; kallikrein inhibitor
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — avoralstat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental): BCX4161 400 mg formulated as hard gelatin capsules given orally under fasting conditions x1
  Interventions: Drug: BCX4161
- Treatment B (Experimental): BCX4161 400 mg formulated as soft gelatin capsules given orally under fasting conditions x1
  Interventions: Drug: BCX4161
- Treatment C (Experimental): BCX4161 400 mg formulated as soft gelatin capsules given orally after a high-fat breakfast x1
  Interventions: Drug: BCX4161

INTERVENTIONS:
Drug: BCX4161 — Each subject will receive Treatments A, B, and C in an open-label, randomized sequence with a washout period of at least 7 days between each dose

SUMMARY:
The purpose of the study is to compare how the body takes up and then eliminates the study drug BCX4161 when it is taken orally as a hard gelatin capsule and as a soft gelatin capsule. This study will also evaluate whether food has any effect on how the body takes up BCX4161.

ELIGIBILITY:
Key Inclusion Criteria:

* Written informed consent
* Body mass index 19 to 32 kg/m2 and a weight of at least 50 kg
* Abide by study restrictions
* Attend all study visits
* Acceptable birth control measures

Key Exclusion Criteria:

* Clinically significant medical history, current medical or psychiatric condition, ECG finding, or laboratory/urinalysis abnormality
* Activated partial thromboplastin time or prothrombin time outside of normal laboratory limits
* Pregnant or nursing
* Recent history of alcohol abuse or positive drugs of abuse screen
* Current smokers
* Donation or loss of greater than 400 mL of blood within 3 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2014-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetics to assess the relative bioavailability of BCX4161 soft gelatin capsules to hard gelatin capsules | Pharmacokinetic parameters AUC0-inf, AUC0-t and Cmax generated after 24 hours of postdose blood sampling

SECONDARY OUTCOMES:
Safety and tolerability evaluated through assessments of adverse events, laboratory analyses, vital signs, ECGs, and physical examinations | Screening through study completion (approximately 61 days)
Plasma pharmacokinetics to assess the effect of food on BCX4161 | Pharmacokinetic parameters AUC0-inf, AUC0-t and Cmax generated after 24 hours of postdose blood sampling

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Collier, Principal Investigator — Quotient Clinical Ltd
Locations (1):
- Quotient Clinical Ltd, Ruddington, Nottingham, United Kingdom